CLINICAL TRIAL: NCT06990646
Title: VR-ACT After Stroke: a Feasibility RCT of a Virtual Reality Delivery of ACT for Pain Management and Mental Health in Patients With Chronic Post-Stroke Pain
Brief Title: VR-ACT After Stroke: a Feasibility Study
Acronym: VR-ACT
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Coimbra (Other)
Collaborators: Unidade Local de Saúde de Coimbra, EPE (Other)
Responsible Party: Principal Investigator, Sérgio Andrade Carvalho, Doctor, University of Coimbra
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 2023.13402.PEX; 2023.13402.PEX (Other Grant/Funding Number: Fundação para a Ciência e Tecnologia (FCT))
Record Dates: First submitted 2025-05-09; First posted 2025-05-25 (Actual); Last update posted 2025-05-25 (Actual); Status verified 2025-05

CONDITIONS: Chronic Pain; Stroke
Keywords: chronic post-stroke pain; contextual-behavioral approaches; virtual reality; acceptance and commitment therapy
MeSH Terms: conditions — Chronic Pain; Stroke

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- VR-ACT (Experimental): 8 modules of 3D immersive skills training (2 targeting awareness regulation skills; 3 promoting acceptance; 3 focused on behavioral change and commitment to valued action)
  Interventions: Behavioral: VR-ACT
- Sham-VR (Sham Comparator): 8 2D non-immersive distracting video animations delivered through a VR headset
  Interventions: Behavioral: Sham-VR

INTERVENTIONS:
Behavioral: VR-ACT — 8 MODULES OF 3D VIRTUAL REALITY Modules 1 & 2: Awareness Regulation Skills Modules 3, 4 & 5: Acceptance of Pain and Internal Experiences Modules 6, 7 & 8: Behavior Change and Valued Action
  Arms: VR-ACT
Behavioral: Sham-VR — 8 2D non-immersive distracting video-animations delivered through a VR headset.
  Arms: Sham-VR

SUMMARY:
This exploratory project aims to develop and pilot test, in a parallel group randomized controlled trial (RCT) design, the feasibility, acceptability, and preliminary efficacy of a self-management virtual reality (VR) 8-week program for pain management and mental health in patients with chronic post-stroke pain (CPSP), in two assessment moments (pre- to post-intervention).

DETAILED DESCRIPTION:
This project has three objectives: O1) to develop and test the feasibility and acceptability of a 8-week VR ACT program (VR-ACT) in a sample of CPSP patients; O2) to pilot test the efficacy of VR-ACT in improving pain, mental health, and adaptive psychological processes and skills, and in reducing the functional connectivity of the Triple Network (DMN, SN, and FPN); O3) To examine the cost-effectiveness of the VR-ACT. The current project will conduct a parallel group design Randomized Controlled Trial (RCT) and will follow a multi-method approach (qualitative and quantitative assessment).

ELIGIBILITY:
Inclusion Criteria:

* medical diagnosis of CPSP;
* age between 18 and 80;
* implicit de facto internet and computer literacy;
* willingness to comply with the study procedures.

Exclusion Criteria:

* currently with active malignancy; -
* severe cognitive impairment;
* currently undergoing any psychological intervention or VR-delivered pain management program;
* current severe psychiatric symptoms (i.e., psychosis; severe depression; non-suicidal self-injury; suicide attempt in the last month);
* language impairment with severe comprehension deficit;
* history of photosensitive epilepsy or previous experience of severe simulator sickness;
* other neurological conditions (e.g., dementia; Parkinson´s).

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-11 (Estimated); Primary Completion 2026-03 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Pain intensity | From enrollment to the end of treatment at 8 weeks
  - The Numeric Rating Scale (NRS)
Pain Impact | From enrollment to the end of treatment at 8 weeks
  - Pain Disability Index (PDI)
Mental Health | From enrollment to the end of treatment at 8 weeks
  Mental Health:
  - Depression Anxiety and Stress Scale (DASS-21)
Psychological and Physical Quality of Life | From enrollment to the end of treatment at 8 weeks
  - World Health Organization Quality of Life - Bref (WHOQOL- Bref)

SECONDARY OUTCOMES:
Mindful Awareness | From enrollment to the end of treatment at 8 weeks
  Mindful Awareness:
  - Mindful Attention Awareness Scale (MAAS)
Emotional Regulation | From enrollment to the end of treatment at 8 weeks
  Emotional Regulation:
  - Difficulties in Emotion Regulation Scale - Short Form (DERS-SF)
Psychological Flexibility | From enrollment to the end of treatment at 8 weeks
  Psychological Flexibility:
  - Comprehensive Assessment of Acceptance and Commitment Therapy Processes (CompACT)

IPD SHARING:
Plan to Share IPD: No